CLINICAL TRIAL: NCT03457701
Title: A Repeat Dose, Open Label, Two Period, Randomized, Cross Over Study to Compare the Effect of Daprodustat to Recombinant, Human Erythropoietin (rhEPO) on Oral Iron Absorption in Adult Participants With Anemia Associated With Chronic Kidney Disease Who Are Not on Dialysis
Brief Title: Anemia Studies in CKD: Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor (PHI) Daprodustat- Iron (ASCEND: Fe)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201771
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Anaemia
Keywords: Recombinant human erythropoietin; Anemia; Daprodustat; Chronic kidney disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned either to remain on their current therapy (either epoetin alfa or darbepoetin alfa) or be switched to daprodustat in either of the treatment periods.
Masking Description: This is an Open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- rhEPO+57Fe followed by Daprodustat+58Fe (Experimental): Participants will be randomly assigned to remain on their current therapy (either epoetin alfa or darbepoetin alfa) in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants will be administered ferrous sulfate containing a stable isotope of iron (57Fe) orally in a randomized fashion following 2 weeks of administration of randomized study treatment. At Day 29 participants will be crossed over to receive Daprodustat in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants will again be administered ferrous sulfate containing the stable iron isotope (58Fe) orally. Participants will be advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: Histamine [H2] receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
  Interventions: Drug: Daprodustat; Drug: rhEPO; Drug: Ferrous sulfate containing the stable iron isotope (57Fe); Drug: Ferrous sulfate containing the stable iron isotope (58Fe)
- rhEPO+58Fe followed by Daprodustat+57Fe (Experimental): Participants will be randomly assigned to remain on their current therapy (either epoetin alfa or darbepoetin alfa) in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants will be administered ferrous sulfate containing a stable isotope of iron (58Fe) orally in a randomized fashion following 2 weeks of administration of randomized study treatment. At Day 29 participants will be crossed over to receive Daprodustat in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants will again be administered ferrous sulfate containing the stable iron isotope (57Fe) orally. Participants will be advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
  Interventions: Drug: Daprodustat; Drug: rhEPO; Drug: Ferrous sulfate containing the stable iron isotope (57Fe); Drug: Ferrous sulfate containing the stable iron isotope (58Fe)
- Daprodustat+57Fe followed by rhEPO+58Fe (Experimental): Participants will be randomly assigned to receive Daprodustat in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants will be administered ferrous sulfate containing a stable isotope of iron (57Fe) orally in a randomized fashion following 2 weeks of administration of randomized study treatment. At Day 29 participants will be crossed over to receive rhEPO (either epoetin alfa or darbepoetin alfa) in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants will again be administered ferrous sulfate containing the stable iron isotope (58Fe) orally. Participants will be advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
  Interventions: Drug: Daprodustat; Drug: rhEPO; Drug: Ferrous sulfate containing the stable iron isotope (57Fe); Drug: Ferrous sulfate containing the stable iron isotope (58Fe)
- Daprodustat+58Fe followed by rhEPO+57Fe (Experimental): Participants will be randomly assigned to receive Daprodustat in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants will be administered ferrous sulfate containing a stable isotope of iron (58Fe) orally in a randomized fashion following 2 weeks of administration of randomized study treatment. At Day 29 participants will be crossed over to receive rhEPO (either epoetin alfa or darbepoetin alfa) in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants will again be administered ferrous sulfate containing the stable iron isotope (57Fe) orally. Participants will be advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
  Interventions: Drug: Daprodustat; Drug: rhEPO; Drug: Ferrous sulfate containing the stable iron isotope (57Fe); Drug: Ferrous sulfate containing the stable iron isotope (58Fe)

INTERVENTIONS:
Drug: Daprodustat — Daprodustat will be available as 1 milligram (mg), 2 mg and 4 mg tablets strengths. One tablet to be taken daily without regard for food.
Drug: rhEPO — rhEPO (epoetin alfa OR darbepoetin alfa) is commercially available in various single dose vials and single-dose prefilled syringes. It will be given as subcutaneous injection.
Drug: Ferrous sulfate containing the stable iron isotope (57Fe) — 57Fe will be available in oral solution. An oral solution will be administered containing 10 mg of 57Fe as ferrous sulfate.
Drug: Ferrous sulfate containing the stable iron isotope (58Fe) — 58Fe will be available in oral solution. An oral solution will be administered containing 3 mg of 58Fe as ferrous sulfate with 7 mg of 56Fe as ferrous sulfate (natural abundance Fe).

SUMMARY:
Daprodustat administration has the potential, by virtue of increasing hypoxia-inducible factor (HIF) levels, to increase oral iron absorption and incorporation into hemoglobin (Hgb). Therefore, the purpose of this study is to compare the effect of daprodustat to rhEPO (i.e., epoetin alfa or darbepoetin alfa) on non-heme oral iron absorption using stable isotopic iron (57Fe and 58Fe) by measuring incorporation of iron in erythrocytes. This study will be a randomized, repeat dose, open label, two period cross-over study in adult, male and female participants with anemia associated with chronic kidney disease who are not on dialysis currently treated with stable doses less than or equal to (<=) 50 percent (%) change in 4-weekly dose) for at least 8 weeks prior to and including the screening period, of rhEPO (i.e., epoetin alfa or darbepoetin alfa). Sufficient participants will be enrolled such that at least 12 participants comprise the Evaluable Population. The study will compare the fractional iron absorption between treatment arms (daprodustat and rhEPO [i.e., epoetin alfa or darbepoetin alfa]) and will evaluate the difference is equal/not equal to zero.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Participants who are Stage 3, 4 or 5 Chronic kidney disease (CKD) (confirmed at Week-4 only) defined by estimated glomerular filtration rate (eGFR) using the CKD Epidemiology Collaboration (CKD-EPI) formula.
* Participants who are currently treated with stable doses (<=50% change in 4-weekly dose) for at least 8 weeks prior to and including the screening period, of rhEPO (i.e., epoetin alfa or darbepoetin alfa).
* Participants with Hgb levels between 9.0 and 11.5 g/dL, inclusive, who meet the Hgb stability criteria.
* Participants may be on stable maintenance oral iron supplementation (less than [<] 50% change in overall dose and compliance of 80% of prescribed doses in the 4 weeks prior to and including the screening period). If participants have been on intravenous (IV) iron, then participants will not have received IV iron for 8 weeks prior to the Day 1 visit.
* Male or Female participants may participate. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP), or a WOCBP who agrees to follow the contraceptive guidance during the treatment period to the follow-up visit.
* Capable of giving signed informed consent.

Exclusion Criteria:

* On dialysis or clinical evidence of impending need to initiate dialysis within 90 days after study start (i.e., Day 1).
* Planned kidney transplant within 3 months after study start.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational products
* Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from screening until the end of Treatment Period 2.
* Planned or current administration of methoxy polyethylene glycol (PEG)-epoetin beta.
* The participant has participated in a clinical trial and has received an experimental investigational product within the prior 30 days or 5 half lives, whichever is longer, from screening through Day 1.
* At or below the lower limit of the reference range at screening for Vitamin B12 (may rescreen in a minimum of 8 weeks).
* Ferritin outside the range between 100 and 500 nanogram per milliliter (ng/mL), inclusive, at screening.
* Transferrin saturation (TSAT) outside the range between 15% and 40%, inclusive, at Screening.
* Folate < 2.0 ng/mL (4.5 nanomoles per liter [nmol/L]; may rescreen in a minimum of 8 weeks) at screening.
* High sensitivity C-reactive protein (hsCRP) >=20 microgram per milliliter (μg/mL) at screening.
* Myocardial infarction or acute coronary syndrome: <=8 weeks prior to screening through Day 1.
* Hospitalization for greater than 24 hours: <=8 weeks prior to screening through Day 1
* Stroke or transient ischemic attack <=8 weeks prior to screening through Day 1.
* Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Current uncontrolled hypertension as determined by the investigator.
* QT interval corrected for heart rate using Bazett's formula (QTcB): QTcB >500 milliseconds (msec), or QTcB > 530 msec in participants with Bundle Branch Block. There is no corrected QT interval (QTc) exclusion for participants with a predominantly paced rhythm.
* Active chronic inflammatory disease that could impact erythropoiesis.
* History of bone marrow aplasia or pure red cell aplasia.
* Conditions, other than anemia associated with chronic kidney disease, which can affect erythropoiesis.
* Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease OR clinically significant gastrointestinal (GI) bleeding from <=4 weeks prior to screening through Day 1.
* Liver disease (any of the following): Alanine transaminase (ALT) >2 times upper limit of normal (ULN; screening only); Bilirubin >1.5 times ULN (screening only). Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Major surgery (excluding vascular access surgery) within the 8 weeks prior to screening through Day 1, or planned during the study.
* Blood transfusion within 8 weeks prior to screening through Day 1, or an anticipated need for blood transfusion during the study.
* Clinical evidence of an acute infection, or history of infection requiring IV antibiotic therapy from 4 weeks prior to screening through Day 1.
* History of malignancy within the two years prior to screening through Day 1 or currently receiving treatment for cancer, with the exception of localized squamous cell or basal cell carcinoma of the skin definitively treated 12 weeks prior to Day 1.
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the participant at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months .
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-period cross over study to compare the effect of Daprodustat to recombinant, human erythropoietin (rhEPO) on oral iron absorption.
Pre-assignment Details: A total of 15 participants were randomized in the study. The safety population consisted of 14 participants who received at least 1 dose of study treatment.
Groups:
- Daprodustat Followed by rhEPO: Participants were randomly assigned to receive Daprodustat in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants were administered ferrous sulfate containing a stable isotope of iron (57Fe or 58Fe) in a randomized fashion following 2 weeks of administration of study treatment. At Day 29 participants were crossed over to receive rhEPO (either epoetin alfa or darbepoetin alfa) in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants were again administered ferrous sulfate containing the stable iron isotope (58Fe or 57Fe). Participants were advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency. There was no washout period between Treatment Period 1 and Treatment Period 2.
- rhEPO Followed by Daprodustat: Participants were randomly assigned to receive rhEPO (i.e., epoetin alfa or darbepoetin alfa) in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants were administered ferrous sulfate containing a stable isotope of iron (57Fe or 58Fe) in a randomized fashion following 2 weeks of administration of study treatment. At Day 29 participants were crossed over to receive Daprodustat in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants were again administered ferrous sulfate containing the stable iron isotope (58Fe or 57Fe). Participants were advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: Histamine [H2] receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency. There was no washout period between Treatment Period 1 and Treatment Period 2.
Period: Treatment Period 1 (up to Day 28)
Arm/Group | Daprodustat Followed by rhEPO | rhEPO Followed by Daprodustat
Started (Randomized) | 7 | 8
Safety Population | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 1
Not completed — Participant reached protocol-defined stopping criteria | 1 | 1
Period: Treatment Period 2 (Up to Day 28)
Arm/Group | Daprodustat Followed by rhEPO | rhEPO Followed by Daprodustat
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Participant reached protocol-defined stopping criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population comprised of participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat Followed by rhEPO | rhEPO Followed by Daprodustat | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (5.35) | 64.6 (13.88) | 65.4 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian/European Heritage | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Fractional Oral Iron Absorption Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected at indicated time points for analysis of fractional oral iron absorption following treatment with Daprodustat and rhEPO. Adjusted mean and 95 percent (%) confidence interval (CI) has been presented.
Time Frame: Up to Day 57
Population: Evaluable Population consisted of all randomized participants who received study medication and completed the iron absorption assessment for both treatment periods.
Measure: Mean (95% Confidence Interval); unit: Percentage (%) of iron absorbed
Groups:
- Daprodustat: Participants were randomly assigned to receive Daprodustat in Treatment Period 1 or 2. For assessment of incorporation of iron into erythrocytes, participants were administered ferrous sulfate containing a stable isotope of iron (57Fe or 58Fe) in a randomized fashion following 2 weeks of administration of study treatment. There was no washout period between treatment periods.
- rhEPO: Participants were randomly assigned to receive rhEPO (i.e., epoetin alfa or darbepoetin alfa) in Treatment Period 1 or 2. For assessment of incorporation of iron into erythrocytes, participants were administered ferrous sulfate containing a stable isotope of iron (57Fe or 58Fe) in a randomized fashion following 2 weeks of administration of study treatment. There was no washout period between treatment periods.
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Percentage (%) of iron absorbed | 20.64 [10.96 to 30.32] | 20.62 [10.95 to 30.30]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; The null hypotheses is defined as the difference in fractional iron absorption between treatment arms (Daprodustat - rhEPO [i.e., epoetin alfa or darbepoetin alfa]) is equal to zero; Test type: Superiority; p = 0.9971, Mixed Models Analysis; Adjusted mean difference. = 0.02, 95% CI 2-sided [-10.13 to 10.16] — Analysis was based on a mixed effects model fitted with fixed effect terms for treatment, period, and iron isotope type and a random participant effect

2. Secondary Outcome: Periods 1 and 2: Change From Baseline in Serum Iron Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected for measurement of serum iron at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: Evaluable Population that included all randomized participants who received study medication and completed the iron absorption assessment for both treatment periods. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Micromoles per liter (umol/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | -1.5 (6.72) | 1.7 (4.93)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 2.5 (8.96) | 3.3 (5.47)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -1.3 (4.93) | -3.5 (6.66)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | -2.2 (4.79) | -3.3 (5.01)

3. Secondary Outcome: Period 1 and 2: Change From Baseline in Transferrin Following Treatment With Daprodustat or rhEPO
Description: Blood samples were collected from participants for measurement of transferrin at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram per Liter (g/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Gram per Liter (g/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.182 (0.2914) | 0.145 (0.2501)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 0.283 (0.2824) | -0.040 (0.1756)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -0.177 (0.4664) | -0.163 (0.2461)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 0.138 (0.2381) | -0.352 (0.2531)

4. Secondary Outcome: Periods 1 and 2: Change From Baseline in Transferrin Saturation Following Treatment With Daprodustat or rhEPO
Description: Blood samples were collected from participants for measurement of transferrin saturation at indicated time points. Transferrin saturation was measured as a percentage and is the ratio of serum iron and total iron-binding capacity multiplied by 100. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of transferrin saturation
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Percentage (%) of transferrin saturation
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | -5.2 (13.63) | 3.5 (12.05)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 3.0 (18.13) | 8.2 (14.41)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -5.5 (13.40) | -4.8 (10.98)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | -6.7 (14.57) | -4.7 (11.29)

5. Secondary Outcome: Periods 1 and 2: Change From Baseline in Soluble Transferrin Receptor Following Treatment of Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of soluble transferrin receptor at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Milligrams per liter (mg/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | -0.218 (0.1736) | 0.063 (0.1669)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | -0.340 (0.2665) | -0.015 (0.1598)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -0.338 (0.2978) | 0.227 (0.1086)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | -0.308 (0.3180) | 0.195 (0.2239)

6. Secondary Outcome: Periods 1 and 2: Ratio to Baseline in Ferritin Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of ferritin at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. The summary of log transformed ration to baseline on markers of iron status for Ferritin is presented here.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per liter (ug/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Microgram per liter (ug/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 1.126 (20.1853) | 0.937 (16.2891)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 1.109 (24.7052) | 1.004 (5.4818)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | 1.067 (32.7697) | 0.957 (20.2623)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 1.278 (53.1128) | 0.911 (23.5414)

7. Secondary Outcome: Periods 1 and 2: Ratio to Baseline (Day 1) in Hepcidin Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of hepcidin at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. The summary of log transformed ration to baseline on markers of iron status for Hepcidin is presented here.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per liter (ug/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Microgram per liter (ug/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.860 (86.4844) | 0.904 (52.1384)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 0.916 (61.2898) | 1.052 (27.7868)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | 0.703 (74.4694) | 1.201 (63.6067)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 0.802 (73.5598) | 1.306 (47.6931)

8. Secondary Outcome: Periods 1 and 2: Change From Baseline in Erythroferrone Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of erythroferrone at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Microgram per liter (ug/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.135 (0.3086) | -0.062 (0.1824)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 0.075 (0.2544) | -0.090 (0.1380)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | 0.063 (0.2225) | -0.068 (0.2405)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 0.032 (0.3578) | -0.110 (0.2278)

9. Secondary Outcome: Periods 1 and 2: Change From Baseline in Hemoglobin Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of hemoglobin at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Grams per liter (g/L)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.7 (3.67) | 2.8 (2.99)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | -5.0 (5.87) | 3.5 (3.39)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -5.3 (4.80) | 3.7 (3.01)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | -4.3 (10.19) | 2.3 (2.94)

10. Secondary Outcome: Periods 1 and 2: Change From Baseline in Hematocrit Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of hematocrit at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Proportion of red blood cells in blood
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.002 (0.0086) | 0.011 (0.0144)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | -0.017 (0.0183) | 0.009 (0.0139)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -0.006 (0.0205) | 0.009 (0.0105)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | -0.010 (0.0343) | 0.002 (0.0114)

11. Secondary Outcome: Periods 1 and 2: Change From Baseline in Erythrocytes Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of erythrocytes (red blood cells number) at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
10^12 cells/liter
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.05 (0.138) | 0.13 (0.137)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | -0.13 (0.163) | 0.13 (0.082)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | -0.17 (0.225) | 0.13 (0.121)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | -0.13 (0.367) | 0.07 (0.151)

12. Secondary Outcome: Periods 1 and 2: Change From Baseline in Erythrocyte Mean Corpuscular Volume Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of erythrocyte mean corpuscular volume at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Femtoliter (fL)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | -0.8 (3.25) | -0.5 (2.43)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | -1.5 (3.45) | -0.8 (2.71)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | 2.8 (4.17) | -0.3 (3.72)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 0.3 (1.97) | -0.8 (3.31)

13. Secondary Outcome: Periods 1 and 2: Change From Baseline in Reticulocyte Hemoglobin Following Treatment of Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of reticulocyte hemoglobin at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
Picogram (pg)
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.333 (1.4334) | -0.033 (0.5888)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 0.250 (1.3925) | 0.717 (0.6882)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | 0.817 (1.5433) | -0.350 (0.7450)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 1.083 (0.8819) | -0.117 (0.9948)

14. Secondary Outcome: Periods 1 and 2: Change From Baseline in Reticulocytes Following Treatment With Daprodustat and rhEPO
Description: Blood samples were collected from participants for measurement of reticulocytes number at indicated time points. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits in the associated treatment period. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Day 14 and Day 28 in treatment periods 1 and 2 (each period is of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 12 | 12
10^12 cells/liter
  Period 1, DAY 14: number analyzed (Participants) | 6 | 6
  Period 1, DAY 14 | 0.001 (0.0155) | 0.002 (0.0090)
  Period 1, DAY 28: number analyzed (Participants) | 6 | 6
  Period 1, DAY 28 | 0.004 (0.0169) | -0.004 (0.0135)
  Period 2, DAY 14: number analyzed (Participants) | 6 | 6
  Period 2, DAY 14 | 0.004 (0.0088) | -0.005 (0.0216)
  Period 2, DAY 28: number analyzed (Participants) | 6 | 6
  Period 2, DAY 28 | 0.020 (0.0099) | -0.010 (0.0213)

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-serious AEs were collected up to Day 73
Description: Safety population comprised of all randomized participants who received at least one dose of study treatment. AEs were presented treatment wise. Participants were followed up for ±3 days following the final sample for assessment of red blood cell iron.
Groups:
- Daprodustat in Period 1: Participants were randomly assigned to receive Daprodustat in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants were administered ferrous sulfate containing a stable isotope of iron (57Fe or 58Fe) in a randomized fashion following 2 weeks of administration of randomized study treatment. Participants were advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
- rhEPO in Period 1: Participants were randomly assigned to receive rhEPO (i.e., epoetin alfa or darbepoetin alfa) in Treatment Period 1. For assessment of incorporation of iron into erythrocytes, participants were administered ferrous sulfate containing a stable isotope of iron (57Fe or 58Fe) in a randomized fashion following 2 weeks of administration of randomized study treatment. Participants were advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: Histamine [H2] receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
- rhEPO in Period 2: At Day 29 participants were crossed over to receive rhEPO (i.e., epoetin alfa or darbepoetin alfa) in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants were again administered ferrous sulfate containing the stable iron isotope (58Fe or 57Fe). Participants were advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
- Daprodustat in Period 2: At Day 29 participants were crossed over to receive Daprodustat in Treatment Period 2. At 2 weeks following initiation of dosing in Treatment Period 2, participants were again administered ferrous sulfate containing the stable iron isotope (58Fe or 57Fe). Participants were advised to maintain use of oral iron supplementation (except ferric citrate) and acid-reducing agents (example: H2 receptor antagonists, proton pump inhibitors, antacids) at a consistent dosage and frequency.
Arm/Group | Daprodustat in Period 1 | rhEPO in Period 1 | rhEPO in Period 2 | Daprodustat in Period 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 3/7 | 3/7 | 2/7 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat in Period 1 (N=7) | rhEPO in Period 1 (N=7) | rhEPO in Period 2 (N=7) | Daprodustat in Period 2 (N=7)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat in Period 1 (N=7) | rhEPO in Period 1 (N=7) | rhEPO in Period 2 (N=7) | Daprodustat in Period 2 (N=7)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT03457701/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT03457701/SAP_001.pdf